CLINICAL TRIAL: NCT00683735
Title: Quantification of the DPP-4 Inhibition-mediated Enhancement of the Activity of the Entero-insular Axis
Brief Title: Quantification of the Dipeptidyl Peptidase (DPP)-4 Inhibition-mediated Enhancement of the Activity of the Entero-insular Axis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Michael A. Nauck (Other)
Responsible Party: Sponsor-Investigator, Michael A. Nauck, Prof. Dr. med., Diabeteszentrum Bad Lauterberg im Harz
Organization: Diabeteszentrum Bad Lauterberg im Harz (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DZBL 2008-Nauck-01; EudraCT: 2008-001663-11
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Diabetes
Keywords: Incretin, DPP-4, metformin, sitagliptin, insulin secretion
MeSH Terms: conditions — Diabetes Mellitus | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Treatment A (Active Comparator): sitagliptin and placebo
  Interventions: Drug: Sitagliptin; Drug: Placebo
- Treatment B (Active Comparator): placebo and metformin
  Interventions: Drug: Metformin; Drug: Placebo
- Treatment C (Active Comparator): sitagliptin and metformin
  Interventions: Drug: Sitagliptin; Drug: Metformin
- Treatment D (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — 100 mg once daily in the morning
  Arms: Treatment A; Treatment C
Drug: Metformin — up to 2000 mg/day
  Arms: Treatment B; Treatment C
Drug: Placebo — 500mg 1-0-0-0
  Arms: Treatment A; Treatment D
Drug: Placebo — 100mg 1-0-0-0
  Arms: Treatment B; Treatment D

SUMMARY:
Objective: To assess the effect if co-administration of sitagliptin and metformin compared to placebo on the incretin effect (based on the comparison of the insulin secretory response to oral glucose load and an 'isoglycaemic' intravenous glucose load). Hypothesis: Treatment with co-administration of sitagliptin and metformin provides a greater incretin effect compared to placebo.

DETAILED DESCRIPTION:
A new class of antidiabetic agents, the DPP-4 inhibitors, are thought to protect endogenously secreted incretin hormones (e.g., GLP-1 and GIP) from proteolytic degradation and inactivation. Since GLP-1 has antidiabetogenic properties, an augmentation of meal-related responses of intact, biologically active GLP-1 can be expected to increase the impact of incretin stimulation to insulin secretory responses. The incretin effect in type 2 diabetic patients is reduced due to an impaired secretion of GLP-1 and a reduced insulinotropic effectiveness of GIP. Therefore, sitagliptin (DPP-4 inhibitor) will be studied in 20 type 2-diabetic patients, who will be treated sequentially (crossover design) with (a) placebo, (b) metformin alone, (c) Sitagliptin alone, and (d) a combination of metformin and Sitagliptin for periods of 6 days (with a washout period of 3 days between treatment. The insulin secretory response (insulin, C-peptide, insulin secretion rates determined by deconvolution analysis) will be compared between experiments with oral glucose (75 g) and "isoglycaemic" intravenous glucose infusions (20% glucose i.v.). The difference represents the "incretin effect". It is expected that the incretin effect in type 2-diabetic patients will be enhanced with sitagliptin treatment, especially combined with metformin.

A secondary objective is to relate the potential increase in the % incretin contribution to insulin secretory response after oral glucose (incretin effect) to changes in the oral glucose-induced response of intact GLP-1 and GIP (measured by specific RIAs). Thus, it will be established, to which degree sitagliptin acts as an "incretin enhancer" in type 2 diabetic patients.

This study will also determine how the combination of sitagliptin to metformin affects the incretin response and insulin secretory response. Metformin is a standard and widely used antihyperglycemic agent which lowers glycemic levels primarily through suppression of hepatic glucose output and improvement in peripheral insulin resistance, resulting in increased glucose transport and utilization by skeletal muscle. There are data to suggest that metformin increases endogenous GLP-1 levels in response to an oral glucose load in obese humans (1).

Therefore it is of relevance to confirm this novel activity of metformin in patients with type 2 diabetes, and to assess potential functional consequences regarding the incretin effect.

ELIGIBILITY:
Inclusion Criteria:

* Type 2-diabetes mellitus
* BMI 25-35 kg/m2
* HbA1c 6.5%-9% (without OHA medication)
* HbA1c 6%-8.5% (OHA monotherapy with metformin or sulfonylurea)
* Patient understands the study-procedures

Exclusion Criteria:

* Type 1-diabetes mellitus
* C-peptide < 0.7ng/mL (0.23 nmol/L)
* Patient has been taking oral anti-hyperglycemic agent (OHA) within the prior 12 weeks, except metformin or a sulfonylurea
* Patient has required insulin therapy within the past 12 weeks

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To assess the effect of co-administration of sitagliptin and metformin compared to placebo on the incretin effect (based on the comparison of the insulin secretory response to oral glucose load and an 'isoglycaemic' intravenous glucose load) | 24 weeks

SECONDARY OUTCOMES:
To assess the effect of sitagliptin compared with placebo on the incretin effect (based on the comparison of the insulin secretory response to oral glucose load and an 'isoglycaemic' intravenous glucose load) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Nauck, Prof. Dr., Principal Investigator — Diabeteszentrum Bad Lauterberg
Locations (1):
- Diabeteszentrum Bad Lauterberg, Bad Lauterberg im Harz, Germany